CLINICAL TRIAL: NCT07002255
Title: A Clinical Study of the Interactions Between Azvudine Tablets (FNC) and Rifampicin Capsules (RIF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GQ-FNC-109
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Azvudine
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : FNC+RIF;RIF;FNC (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Rifampicin Capsules (RIF)
- Group 2 : FNC;FNC+RIF;RIF (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Rifampicin Capsules (RIF)
- Group 3 : RIF;FNC;FNC+RIF (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Rifampicin Capsules (RIF)

INTERVENTIONS:
Drug: Azvudine tablets(FNC) and Rifampicin Capsules (RIF) — This study consisted of 3 cycles, each cycle was administered orally for 7 consecutive days, and the washout period between each cycle was 7 days. Subjects were administered the drug as follow:
  FNC 3mg (1 tablet)+RIF 600 mg (4 capsules) (taken at the same time), 1 time a day, orally, for 7 consecutive days; RIF: 600 mg (4 capsules) each time, 1 time a day, orally, for 7 consecutive days; FNC: 3 mg (1 tablet) each time, 1 time a day, orally, for 7 consecutive days.
  Arms: Group 1 : FNC+RIF;RIF;FNC
Drug: Azvudine tablets(FNC) and Rifampicin Capsules (RIF) — This study consisted of 3 cycles, each cycle was administered orally for 7 consecutive days, and the washout period between each cycle was 10 days. Subjects were administered the drug as follow:
  FNC: 3 mg (1 tablet) each time, 1 time a day, orally, for 7 consecutive days; FNC 3mg (1 tablet) +RIF 600 mg (4 capsules) (taken at the same time), 1 time a day, orally, for 7 consecutive days; RIF: 600 mg (4 capsules) each time, 1 time a day, orally, for 7 consecutive days.
  Arms: Group 2 : FNC;FNC+RIF;RIF
Drug: Azvudine tablets(FNC) and Rifampicin Capsules (RIF) — This study consisted of 3 cycles, each cycle was administered orally for 7 consecutive days, and the washout period between each cycle was 10 days. Subjects were administered the drug as follow:
  RIF: 600 mg (4 capsules), 1 time a day, orally, for 7 consecutive days; FNC: 3 mg (1 tablet) each time, 1 time a day, orally, for 7 consecutive days; FNC 3mg (1 tablet)+RIF 600 mg (4 capsules) (taken at the same time), 1 time a day, orally, for 7 consecutive days.
  Arms: Group 3 : RIF;FNC;FNC+RIF

SUMMARY:
Azvudine(FNC)，a nucleoside reverse transcriptase inhibitor, make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance. FNC is a broad-spectrum RNA virus inhibitor that inhibits the novel coronavirus RNA-dependent RNA polymerase (RdRp).

This is a clinical study to evaluate the Interactions between Azvudine Tablets (FNC) and Rifampicin Capsules (RIF) in healthy subjects. This is a single-center, randomized, open-label, three-cycles, three-treatment crossover clinical trial. Subjects was administered orally for 7 consecutive days each cycle, and the washout period between each cycle was 7 days. Biological sample collection and safety examination were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged ≥ 18 years old and ≤ 45 years old, regardless of gender;
2. Body mass index (BMI) within the range of 19.0-26.0 (including the critical value) (BMI = weight (kg) / height 2 (m2)), the weight of men should be ≥ 50.0kg, and the weight of women should be ≥ 45.0kg;
3. Those who had no birth plan within 2 weeks before screening and within 6 months after the end of the trial and agree to take effective non-drug contraceptive measures during the trial;
4. Understand and sign the informed consent form.

Exclusion Criteria:

1. Persons with allergic constitutions, history of drug or food allergies, especially those who were allergic to any ingredient in this product and its excipients;
2. Individuals with a history of hypoglycemia;
3. Individuals deemed ineligible by the clinical research physician due to significant clinical abnormalities in medical history, physical examination, laboratory tests, and other related examinations;
4. Individuals with a history of smoking addiction within 12 months prior to screening (the number of cigarettes smoked ≥5 per day);
5. Individuals with a history of alcohol abuse within the past 12 months (consuming ≥14 units of alcohol weekly: 1 unit = 285 mL of beer, or 25 mL of spirits, or 150 mL of wine), or who tested positive for alcohol on breath tests prior to study enrollment (testing value >0mg/100mL);
6. Individuals with a history of substance abuse within the past 12 months or who tested positive for addictive substances prior to enrollment;
7. Individuals who underwent surgery within the past 3 months, especially those who had had surgeries that would affect drug absorption, distribution, metabolism, or excretion, or those planning to undergo surgery during the study;
8. Individuals who had taken any medication that interacts with the trial drug in the 30 days prior to screening, such as: isoniazid, ethionamide, chlorphenozine, miconazole, ketoconazole, etc.;
9. Individuals with a history of cardiovascular, liver, kidney, pulmonary, gastrointestinal, neurological diseases, especially any surgical conditions or disorders that might affect drug absorption, distribution, metabolism, and excretion, or any surgical conditions or disorders that might pose hazards to participants;
10. Individuals with febrile illness within the 3 days prior to screening;
11. Individuals who had participated in any other clinical trials within the past 3 months;
12. Individuals with any history of prescription drugs, over-the-counter drugs, herbal medicine, or dietary supplements within 14 days prior to screening;
13. Individuals who had been vaccinated against the novel coronavirus within 14 days before screening or other vaccines within 3 months before screening or planed to be vaccinated during the trial;
14. Individuals who had consumed excessive tea, coffee, and/or caffeinated, xanthine, or alcoholic beverages (more than 8 cups, 1 cup = 250 mL) daily within the 3 months prior to screening;
15. Individuals who had lost blood or donated ≥200 mL within the past 8 weeks;
16. Pregnant or breastfeeding women;
17. Individuals who could not tolerate venipuncture or had a history of vasovagal syncope;
18. Individuals deemed unsuitable for this study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration at Steady State (Cmax, ss) of Azvudine and Rifampicin | Blood samples were collected on Day 5, 6, 7, 18, 19, 20, 31, 32 and 33 of the study.
Pharmacokinetics (PK): Time to Maximum Plasma Concentration at Steady State (Tmax, ss) of Azvudine and Rifampicin | Blood samples were collected on Day 5, 6, 7, 18, 19, 20, 31, 32 and 33 of the study.
Pharmacokinetics (PK): Elimination of Terminal Half-Life (t1/2) of Azvudine and Rifampicin | Blood samples were collected on Day 5, 6, 7, 18, 19, 20, 31, 32 and 33 of the study.

SECONDARY OUTCOMES:
Occurrence of Adverse Events | From enrollment to the end of the study on Day 34.
  Clinical presentation characteristics, severity, onset time, duration of adverse events, management measures, outcomes, and the correlation with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Heping Hospital Affliliated to Changzhi Medical College, Shanxi, China